CLINICAL TRIAL: NCT01972438
Title: A Randomized, Controlled, Double-Masked, Clinical Trial of Autologous Serum Eye Drops for Severe Ocular Chronic Graft-versus-Host Disease (GVHD) in Hematopoietic Stem Cell Transplant (HSCT) Patients
Acronym: GVHD ASED
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigational product unavailable due to manufacturing issues
Sponsor: National Eye Institute (NEI) (NIH)
Collaborators: The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 130206; 13-EI-0206
Record Dates: First submitted 2013-10-23; First posted 2013-10-30 (Estimated); Results first posted 2016-09-13 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-10

CONDITIONS: Graft vs Host Disease
Keywords: Graft Versus Host Disease; Hematopoietic Stem Cell Transplant
MeSH Terms: conditions — Graft vs Host Disease | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ASEDs - Saline (Experimental): Participants administer autologous serum eye drops (ASEDs) daily for the first three months, then crossover to administer control (normal saline) eye drops daily beginning at Month 3 through Month 6.
  Interventions: Drug: ASEDs; Drug: Saline
- Saline - ASEDs (Placebo Comparator): Participants administer control (normal saline) eye drops daily for the first three months, then crossover to administer autologous serum eye drops (ASEDs) daily beginning at Month 3 through Month 6.
  Interventions: Drug: ASEDs; Drug: Saline

INTERVENTIONS:
Drug: ASEDs — Experimental Intervention
Drug: Saline — Control Intervention

SUMMARY:
Some eye diseases can be helped by eye drops made from a person's own blood. These eye drops are called autologous serum eye drops, or ASEDs. ASEDs have been studied in only a few people with graft vs. host disease (GVHD) affecting the eye and were found to be helpful with few side effects.

The purpose of this study was to determine whether ASEDs are safe and more effective than control (normal saline) and can help with eye symptoms in people with severe chronic eye GVHD.

Each participant in this study was to have blood drawn to prepare ASEDs specifically for the participant. Each participant was scheduled to receive ASEDs for 3 months and placebo eye drops (salt water) for 3 months. Participants did not know when they were receiving the ASEDs and when they were receiving placebo eye drops.

DETAILED DESCRIPTION:
Objective:

A common, serious and debilitating long term complication of hematopoietic stem cell transplant (HCST) is chronic graft-versus-host disease (GVHD). Ocular GVHD develops in up to 85% of patients with chronic GVHD. It is characterized by progressive keratitis sicca and cicatrizing ocular inflammatory surface disease with T cell mediated damage to conjunctival and corneal epithelium and lacrimal tissue. Various medical and surgical treatments have been used, such as various lubricating agents, steroid drops and ointments, cyclosporin drops, punctal plugs or cautery and partial tarsorrhaphy. However, in severe cases, none offer acceptable, long-lasting relief from pain, irritation, dryness and diminished vision associated with ocular GVHD. An alternative treatment that has previously been safely investigated is autologous serum eye drops (ASEDs). The objective of this study was to determine whether ASEDs are more effective than control (normal saline) in the treatment of severe chronic ocular GVHD in HSCT patients unresponsive to standard medical treatment.

Study Population:

Eighteen post-HSCT patients with severe ocular GVHD unresponsive to standard medical treatment were enrolled. Initially, 34 post-HSCT patients with severe ocular GVHD unresponsive to standard medical treatment were to be enrolled. However, only 18 enrolled, as the investigational product (IP) was no longer provided to participants as of June 2015 due to manufacturing issues.

Design:

This was a Phase 2, randomized, double-masked, controlled, crossover, single-center study to investigate ASEDs in participants with severe chronic ocular GVHD. During the initial crossover phase of the study, participants participated in a two-period, six-month, crossover study in which participants were randomized to one of two treatment sequence groups. The two groups were: 1) daily administration of ASEDs for the first three months and then crossover to control (normal saline) eye drops beginning at Month 3 through Month 6, or 2) daily administration of control (normal saline) eye drops for the first three months and then crossover to ASEDs beginning at Month 3 through Month 6. Participants in both groups applied the assigned drops four times per day for six months, as well as maintained their current standard ocular GVHD therapy. Following the initial crossover phase, beginning at the Month 6 visit, participants were provided ASEDs as open-label treatment on an as-needed basis until study completion. As of June 2015, participants were informed to discontinue use of the IP and send it back the NIH Pharmacy. During the first year, required clinic visits occurred at Baseline, Months 3, 6 and 12 with required telephone follow-up visits at Months 7 and 9. Following the Month 12 visit, participants were evaluated every six months, alternating telephone follow-up visits with clinic visits, until the last enrolled participant reached his/her Month 12 visit. At the discretion of the Investigator, participants who did not complete the Month 12 visit had the most recent study visit constitute as the final safety visit, otherwise the participant was scheduled for a final safety visit within 4 1/2 months. Participants who already surpassed the Month 12 visit were scheduled for a final safety visit within 4 1/2 months.

Outcome Measures:

The primary outcome was the proportion of participants experiencing a ≥ 50% reduction in the combined score of the modified Oxford punctate keratopathy grading and the National Institutes of Health (NIH)/National Eye Institute (NEI) visual analogue scale in the study eye from baseline to Month 3. A ≥ 50% reduction in the combined score is considered a treatment success. While the design is a crossover study, the primary outcome was assessed after the first period at Month 3. Secondary outcomes included changes in the combined score of the modified Oxford punctate keratopathy grading and the NIH/NEI visual analogue scale in both eyes from baseline to the end of each period, changes in the chronic ocular GVHD Composite Assessment Scale (CAS) score, objective testing, subjective testing and global chronic GVHD assessments in both eyes. Safety outcomes were the number and severity of systemic and ocular toxicities and adverse events. The number of participants withdrawn from the study treatment due to vision loss, adverse events or treatment failure also contributed to the assessment of safety.

ELIGIBILITY:
Inclusion Criteria

1. Participant must be 18 years of age or older.
2. Participant must understand and sign the protocol's informed consent document.
3. Participant must have severe ocular Graft-versus-host Disease (GVHD) in one (unilateral) or both (bilateral) eyes with the following characteristics in the study eye:

   1. Combined score of modified Oxford punctate keratopathy grading and National Institutes of Health (NIH)/National Eye Institute (NEI) visual analogue scale of ≥ 4, and
   2. Composite assessment scale (CAS) score of ≥ 3, and
   3. Schirmer's tear test without anesthesia of ≤ 5 mm, and
   4. Not responsive to standard medical treatment for at least three months prior to randomization. Standard medical treatment includes cyclosporine (Restasis®) ophthalmic emulsion (if tolerated), steroid drops (unless contraindicated), lubricating drops and ointments.
4. Participant is enrolled in an NIH study at the National Cancer Institute (NCI) or National Heart, Lung and Blood Institute (NHLBI).
5. Participant is willing and able to supply an adequate amount of blood to create the autologous serum eye drops (ASEDs).

Exclusion Criteria

1. Participant is unable to comply with study procedures or follow-up visits.
2. Participant is seropositive with positive nucleic acid confirmatory tests for human immunodeficiency virus-1/2 (HIV-1/2), human T lymphotropic virus-I/II (HTLV-I/II), hepatitis C virus (HCV), and/or hepatitis B virus (HBV) without confirmed history of vaccination.
3. Participant has GVHD proliferative keratopathy, uveitis or GVHD retinopathy in either eye.
4. Participant has an active ocular infection in either eye.
5. Participant has an allergy to dilating or anesthetic eye drops.
6. Participant has used Boston Scleral Lens (or similar lenses) in either eye or has used ASEDs in either eye within the past two months. Participants who have used the Boston Scleral Lens (or similar lenses) or ASEDs in either eye who did not respond to treatment and have stopped using them for at least two months are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-11; Primary Completion 2015-05 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel B Datiles, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Filipovich AH, Weisdorf D, Pavletic S, Socie G, Wingard JR, Lee SJ, Martin P, Chien J, Przepiorka D, Couriel D, Cowen EW, Dinndorf P, Farrell A, Hartzman R, Henslee-Downey J, Jacobsohn D, McDonald G, Mittleman B, Rizzo JD, Robinson M, Schubert M, Schultz K, Shulman H, Turner M, Vogelsang G, Flowers ME. National Institutes of Health consensus development project on criteria for clinical trials in chronic graft-versus-host disease: I. Diagnosis and staging working group report. Biol Blood Marrow Transplant. 2005 Dec;11(12):945-56. doi: 10.1016/j.bbmt.2005.09.004. PMID 16338616
- [Background] Yamada C, King KE, Ness PM. Autologous serum eyedrops: literature review and implications for transfusion medicine specialists. Transfusion. 2008 Jun;48(6):1245-55. doi: 10.1111/j.1537-2995.2008.01665.x. Epub 2008 Apr 10. PMID 18410252
- [Background] Bron AJ, Evans VE, Smith JA. Grading of corneal and conjunctival staining in the context of other dry eye tests. Cornea. 2003 Oct;22(7):640-50. doi: 10.1097/00003226-200310000-00008. PMID 14508260
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-EI-0206.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Initially, up to 34 participants were to be enrolled. However, due to the unavailability of the investigational product (IP), recruitment and enrollment was halted at 18 participants in May 2015, and the study closed early. Three participants were enrolled and randomized but unrelated to the early study closure never started IP.
Groups:
- ASEDs - Saline: Participants administer autologous serum eye drops (ASEDs) daily for the first three months, then crossover to administer control (normal saline) eye drops daily beginning at Month 3 through Month 6.
  ASEDs - Saline: Experimental Intervention
- Saline - ASEDs: Participants administer control (normal saline) eye drops daily for the first three months, then crossover to administer autologous serum eye drops (ASEDs) daily beginning at Month 3 through Month 6.
  Saline - ASEDs: Control Intervention
Period: Baseline-Month 3 Crossover Period
Arm/Group | ASEDs - Saline | Saline - ASEDs
Started | 9 (Two participants never started IP: one died and one did not meet the inclusion criteria) | 9 (One participant never started IP, as unable to donate blood for preparation of ASEDs)
Completed | 6 | 6
Not Completed | 3 | 3
Not completed — Death | 1 | 0
Not completed — Did not meet inclusion criteria | 1 | 0
Not completed — Unable to donate blood | 0 | 1
Not completed — Scheduling difficulties (Missed Month 3) | 1 | 2
Period: Months 3-6 Crossover Period
Arm/Group | ASEDs - Saline | Saline - ASEDs
Started | 6 | 7 (Two participants who missed Month 3 visit completed this pd but one who completed Month 3 didn't)
Completed | 6 | 6
Not Completed | 0 | 1
Not completed — Early Study Closure | 0 | 1
Period: Months 6-12 Study Period
Arm/Group | ASEDs - Saline | Saline - ASEDs
Started | 6 | 6
Completed | 3 | 4
Not Completed | 3 | 2
Not completed — Death | 1 | 0
Not completed — Early Study Closure | 2 | 2
Period: Post Month 12 Study Period
Arm/Group | ASEDs - Saline | Saline - ASEDs
Started | 3 | 4
Completed | 0 | 0
Not Completed | 3 | 4
Not completed — Early Study Closure | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ASEDs - Saline | Saline - ASEDs | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 6 | 14
  >=65 years | 1 | 3 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.1 (13.49) | 53.4 (14.77) | 49.3 (14.38)
Gender [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 9 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 8 | 8 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Who Experienced a ≥ 50% Reduction in the Combined Score of the Modified Oxford Punctate Keratopathy Grading and the NIH/National Eye Institute (NEI) Visual Analogue Scale in the Study Eye From Baseline to Month 3.
Description: A ≥ 50% reduction in the combined score was considered a treatment success. While the design is a crossover study, the primary outcome was assessed after the first period at Month 3. Oxford punctate keratopathy is an objective measure from 0-5 (cornea only) and the NIH/NEI visual analogue scale is a subjective grading performed by the participant regarding his/her ocular dryness, redness and irritation (scored 0-3 for each symptom with 0 = none, 1 = mild, 2 = moderate and 3 = severe for a total score between 0-9). The combined score was a number between 0-14 with the higher number representing a worse outcome.
Time Frame: Baseline and 3 months
Population: This analysis is conducted on the per-protocol population, defined as those who adhered to the protocol prior to drug unavailability, not on the intent-to-treat population due to lack of visit information beyond baseline for 3 participants. Three never started drug: one was unable to donate blood, one was ineligible at screening and one died.
Measure: Number; unit: participants
Units Other Than Participants: eyes
Arm/Group | ASEDs - Saline | Saline - ASEDs
Number analyzed (Participants) | 6 | 6
Number analyzed (eyes) | 6 | 6
participants | 1 | 0

2. Secondary Outcome: Number of Systemic and Ocular Toxicities and Adverse Events
Time Frame: Study Duration, up to 24 months
Measure: Number; unit: adverse events
Arm/Group | ASEDs - Saline | Saline - ASEDs
Number analyzed (Participants) | 9 | 9
adverse events | 4 | 5

3. Secondary Outcome: Number of Participants Withdrawn From the Study Treatment Due to Vision Loss, Adverse Events or Treatment Failure
Time Frame: Study Duration, up to 24 months
Measure: Number; unit: participants
Arm/Group | ASEDs - Saline | Saline - ASEDs
Number analyzed (Participants) | 9 | 9
participants | 0 | 0

4. Secondary Outcome: Mean Change in the Combined Score of the Modified Oxford Punctate Keratopathy Grading and the NIH Visual Analogue Scale in the Study Eye at 3 Months Compared to Baseline
Description: Oxford punctate keratopathy is an objective measure from 0-5 (cornea only) and the NIH/NEI visual analogue scale is a subjective grading performed by the participant regarding his/her ocular dryness, redness and irritation (scored 0-3 for each symptom with 0 = none, 1 = mild, 2 = moderate and 3 = severe for a total score between 0-9). The combined score was a number between 0-14 with the higher number representing a worse outcome.
Time Frame: Baseline and 3 Months
Population: Twelve participants completed the first crossover treatment period at Month 3.
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: eyes
Arm/Group | ASEDs - Saline | Saline - ASEDs
Number analyzed (Participants) | 6 | 6
Number analyzed (eyes) | 6 | 6
scores on a scale | -4.1 (1.8) | -2.6 (2.8)

5. Secondary Outcome: Mean Change in the Combined Score of the Modified Oxford Punctate Keratopathy Grading and the NIH Visual Analogue Scale in the Fellow Eye at 3 Months Compared to Baseline
Description: The fellow eye is the untreated eye. Oxford punctate keratopathy is an objective measure from 0-5 (cornea only) and the NIH/NEI visual analogue scale is a subjective grading performed by the participant regarding his/her ocular dryness, redness and irritation (scored 0-3 for each symptom with 0 = none, 1 = mild, 2 = moderate and 3 = severe for a total score between 0-9). The combined score was a number between 0-14 with the higher number representing a worse outcome.
Time Frame: Baseline and 3 Months
Population: Twelve participants completed the first crossover treatment period at Month 3.
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: eyes
Arm/Group | ASEDs - Saline | Saline - ASEDs
Number analyzed (Participants) | 6 | 6
Number analyzed (eyes) | 6 | 6
scores on a scale | -2.1 (2.5) | -2.5 (3.5)

6. Secondary Outcome: Mean Change in the Combined Score of the Modified Oxford Punctate Keratopathy Grading and the NIH Visual Analogue Scale in the Study Eye at 6 Months Compared to Baseline
Description: as for outcome 4
Time Frame: Baseline and 6 Months
Population: Twelve participants completed the first crossover treatment period at Month 3. Thirteen participants completed the second crossover treatment period at Month 6.
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: eyes
Arm/Group | ASEDs - Saline | Saline - ASEDs
Number analyzed (Participants) | 7 | 6
Number analyzed (eyes) | 7 | 6
scores on a scale | -4.1 (3.7) | -0.5 (3.0)

7. Secondary Outcome: Mean Change in the Combined Score of the Modified Oxford Punctate Keratopathy Grading and the NIH Visual Analogue Scale in the Fellow Eye at 6 Months Compared to Baseline
Description: as for outcome 5
Time Frame: Baseline and 6 Months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: eyes
Arm/Group | ASEDs - Saline | Saline - ASEDs
Number analyzed (Participants) | 7 | 6
Number analyzed (eyes) | 7 | 6
scores on a scale | -2.4 (2.2) | -2.7 (1.9)

8. Secondary Outcome: Mean Change in the Chronic Ocular GVHD Composite Assessment Scale (CAS) Score in the Study Eye at 3 Months Compared to Baseline
Description: The CAS score is the sum of the scores on three separate assessments: Schirmer's tear test without anesthesia, punctate keratopathy and conjunctival inflammation and scarring (scored according to Robinson et. al*). Each assessment was scored 0-3 with 0 = none, 1 = mild, 2 = moderate and 3 = severe. The higher values represent a worse outcome. The CAS score was a number between 0-9 with the higher number representing a worse outcome.
  *Robinson MR, Lee SS, Rubin BI, Wayne AS, Pavletic SZ, Bishop MR, Childs R, Barrett AJ, Csaky KG. Topical Corticosteroid Therapy for Cicatricial Conjunctivitis Associated with Chronic Graft Versus Host Disease. Bone Marrow Transplant. 2004; 18:567-9.
Time Frame: Baseline and 3 Months
Population: Twelve participants completed the first crossover treatment period at Month 3.
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: eyes
Arm/Group | ASEDs - Saline | Saline - ASEDs
Number analyzed (Participants) | 6 | 6
Number analyzed (eyes) | 6 | 6
scores on a scale | -1.2 (2.3) | -1.0 (1.3)

9. Secondary Outcome: Mean Change in the Chronic Ocular GVHD Composite Assessment Scale (CAS) Score in the Fellow Eye at 3 Months Compared to Baseline
Description: The fellow eye is the untreated eye. The CAS score is the sum of the scores on three separate assessments: Schirmer's tear test without anesthesia, punctate keratopathy and conjunctival inflammation and scarring (scored according to Robinson et. al*). Each assessment was scored 0-3 with 0 = none, 1 = mild, 2 = moderate and 3 = severe. The higher values represent a worse outcome. The CAS score was a number between 0-9 with the higher number representing a worse outcome.
  *Robinson MR, Lee SS, Rubin BI, Wayne AS, Pavletic SZ, Bishop MR, Childs R, Barrett AJ, Csaky KG. Topical Corticosteroid Therapy for Cicatricial Conjunctivitis Associated with Chronic Graft Versus Host Disease. Bone Marrow Transplant. 2004; 18:567-9.
Time Frame: Baseline and 3 Months
Population: Twelve participants completed the first crossover treatment period at Month 3.
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: eyes
Arm/Group | ASEDs - Saline | Saline - ASEDs
Number analyzed (Participants) | 6 | 6
Number analyzed (eyes) | 6 | 6
scores on a scale | 1.5 (7.1) | 0.8 (1.9)

10. Secondary Outcome: Mean Change in the Chronic Ocular GVHD Composite Assessment Scale (CAS) Score in the Study Eye at 6 Months Compared to Baseline
Description: as for outcome 8
Time Frame: Baseline and 6 Months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: eyes
Arm/Group | ASEDs - Saline | Saline - ASEDs
Number analyzed (Participants) | 7 | 6
Number analyzed (eyes) | 7 | 6
scores on a scale | -1.8 (3.1) | -0.4 (2.6)

11. Secondary Outcome: Mean Change in the Chronic Ocular GVHD Composite Assessment Scale (CAS) Score in the Fellow Eye at 6 Months Compared to Baseline
Description: as for outcome 9
Time Frame: Baseline and 6 Months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: eyes
Arm/Group | ASEDs - Saline | Saline - ASEDs
Number analyzed (Participants) | 7 | 6
Number analyzed (eyes) | 7 | 6
scores on a scale | -0.6 (1.8) | -0.2 (5.8)

12. Secondary Outcome: Mean Change in Early Treatment Diabetic Retinopathy Study (ETDRS) Best-corrected Visual Acuity (BCVA) in the Study Eye at 3 Months Compared to Baseline.
Description: Visual acuity was measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol. Acuity is measured as letters read on an ETDRS eye chart and the letters read equate to Snellen measurements. For example, if a participant reads between 84 and 88 letters, the equivalent Snellen measurement is 20/20.
Time Frame: Baseline and 3 Months
Population: Twelve participants completed the first crossover treatment period at Month 3.
Measure: Mean (Standard Deviation); unit: ETDRS letters
Units Other Than Participants: eyes
Arm/Group | ASEDs - Saline | Saline - ASEDs
Number analyzed (Participants) | 6 | 6
Number analyzed (eyes) | 6 | 6
ETDRS letters | -2.3 (4.3) | -7.2 (22.7)

13. Secondary Outcome: Mean Change in Early Treatment Diabetic Retinopathy Study (ETDRS) Best-corrected Visual Acuity (BCVA) in the Fellow Eye at 3 Months Compared to Baseline
Description: The fellow eye is the untreated eye. Visual acuity was measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol. Acuity is measured as letters read on an ETDRS eye chart and the letters read equate to Snellen measurements. For example, if a participant reads between 84 and 88 letters, the equivalent Snellen measurement is 20/20.
Time Frame: Baseline and 3 Months
Population: Twelve participants completed the first crossover treatment period at Month 3.
Measure: Mean (Standard Deviation); unit: ETDRS letters
Units Other Than Participants: eyes
Arm/Group | ASEDs - Saline | Saline - ASEDs
Number analyzed (Participants) | 6 | 6
Number analyzed (eyes) | 6 | 6
ETDRS letters | 1.5 (2.4) | 0.3 (3.5)

14. Secondary Outcome: Mean Change in Early Treatment Diabetic Retinopathy Study (ETDRS) Best-corrected Visual Acuity (BCVA) in the Study Eye at 6 Months Compared to Baseline
Description: as for outcome 12
Time Frame: Baseline and 6 Months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ETDRS letters
Units Other Than Participants: eyes
Arm/Group | ASEDs - Saline | Saline - ASEDs
Number analyzed (Participants) | 7 | 6
Number analyzed (eyes) | 7 | 6
ETDRS letters | 1.8 (8.0) | -4.3 (6.7)

15. Secondary Outcome: Mean Change in Early Treatment Diabetic Retinopathy Study (ETDRS) Best-corrected Visual Acuity (BCVA) in the Fellow Eye at 6 Months Compared to Baseline.
Description: as for outcome 13
Time Frame: Baseline and 6 Months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ETDRS letters
Units Other Than Participants: eyes
Arm/Group | ASEDs - Saline | Saline - ASEDs
Number analyzed (Participants) | 7 | 6
Number analyzed (eyes) | 7 | 6
ETDRS letters | 0.6 (8.6) | -2.2 (6.7)

16. Secondary Outcome: Mean Change in Tear Stability (Tear Break-up Time) in the Study Eye at 3 Months Compared to Baseline
Description: Sodium fluorescein dye was added to the eye and the tear film was observed under the slit lamp while the participant avoided blinking until tiny dry spots develop. Three measurements were taken and averaged for a more reproducible score.
Time Frame: Baseline and 3 Months
Population: Twelve participants completed the first crossover treatment period at Month 3.
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: eyes
Arm/Group | ASEDs - Saline | Saline - ASEDs
Number analyzed (Participants) | 6 | 6
Number analyzed (eyes) | 6 | 6
seconds | 3.7 (6.0) | 1.4 (2.1)

17. Secondary Outcome: Mean Change in Tear Stability (Tear Break-up Time) in the Fellow Eye at 3 Months Compared to Baseline
Description: The fellow eye is the untreated eye. Sodium fluorescein dye was added to the eye and the tear film was observed under the slit lamp while the participant avoided blinking until tiny dry spots develop. Three measurements were taken and averaged for a more reproducible score.
Time Frame: Baseline and 3 Months
Population: Twelve participants completed the first crossover treatment period at Month 3.
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: eyes
Arm/Group | ASEDs - Saline | Saline - ASEDs
Number analyzed (Participants) | 6 | 6
Number analyzed (eyes) | 6 | 6
seconds | 3.3 (5.1) | 2.3 (2.9)

18. Secondary Outcome: Mean Change in Tear Stability (Tear Break-up Time) in the Study Eye at 6 Months Compared to Baseline
Description: as for outcome 16
Time Frame: Baseline and 6 Months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: eyes
Arm/Group | ASEDs - Saline | Saline - ASEDs
Number analyzed (Participants) | 7 | 6
Number analyzed (eyes) | 7 | 6
seconds | 0.2 (1.5) | 0.6 (0.7)

19. Secondary Outcome: Mean Change in Tear Stability (Tear Break-up Time) in the Fellow Eye at 6 Months Compared to Baseline
Description: as for outcome 17
Time Frame: Baseline and 6 Months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: eyes
Arm/Group | ASEDs - Saline | Saline - ASEDs
Number analyzed (Participants) | 7 | 6
Number analyzed (eyes) | 7 | 6
seconds | -0.1 (2.3) | -0.1 (1.3)

20. Secondary Outcome: Mean Change in Tear Composition (Tear Osmolarity) in the Study Eye at 3 Months Compared to Baseline
Description: The tear composition test consists of the measurement of tear osmolarity using the Tearlab Osmolarity System (San Diego, California) by collecting a small 50 nanoliter (nL) tear sample which, with the use of laboratory test calculations, can derive the tear osmolarity in milliosmole per liter (mOsm/L).
Time Frame: Baseline and 3 Months
Population: Twelve participants completed the first crossover treatment period at Month 3.
Measure: Mean (Standard Deviation); unit: mOsm/L
Units Other Than Participants: eyes
Arm/Group | ASEDs - Saline | Saline - ASEDs
Number analyzed (Participants) | 6 | 6
Number analyzed (eyes) | 6 | 6
mOsm/L | 2.3 (20) | -32.8 (24.5)

21. Secondary Outcome: Mean Change in Tear Composition (Tear Osmolarity) in the Study Eye at 6 Months Compared to Baseline
Description: as for outcome 20
Time Frame: Baseline and 6 Months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mOsm/L
Units Other Than Participants: eyes
Arm/Group | ASEDs - Saline | Saline - ASEDs
Number analyzed (Participants) | 7 | 6
Number analyzed (eyes) | 7 | 6
mOsm/L | 13.5 (3.5) | 3.8 (15.9)

22. Secondary Outcome: Mean Change in Tear Composition (Tear Osmolarity) in the Fellow Eye at 3 Months Compared to Baseline
Description: The fellow eye is the untreated eye. The tear composition test consists of the measurement of tear osmolarity using the Tearlab Osmolarity System (San Diego, California) by collecting a small 50 nanoliter (nL) tear sample which, with the use of laboratory test calculations, can derive the tear osmolarity in milliosmole per liter (mOsm/L).
Time Frame: Baseline and 3 Months
Population: Twelve participants completed the first crossover treatment period at Month 3.
Measure: Mean (Standard Deviation); unit: mOsm/L
Units Other Than Participants: eyes
Arm/Group | ASEDs - Saline | Saline - ASEDs
Number analyzed (Participants) | 6 | 6
Number analyzed (eyes) | 6 | 6
mOsm/L | -0.2 (28.5) | -1.3 (12.0)

23. Secondary Outcome: Mean Change in Tear Composition (Tear Osmolarity) in the Fellow Eye at 6 Months Compared to Baseline
Description: as for outcome 22
Time Frame: Baseline and 6 Months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mOsm/L
Units Other Than Participants: eyes
Arm/Group | ASEDs - Saline | Saline - ASEDs
Number analyzed (Participants) | 7 | 6
Number analyzed (eyes) | 7 | 6
mOsm/L | 4.5 (0.7) | 6.0 (37.6)

ADVERSE EVENTS:
Time Frame: Study Duration, up to 24 months
Description: Of the events:1 occurred while participant was taking autologous serum eye drops (ASEDs);3 occurred when participant(s) were taking normal saline eye drops;3 occurred prior to starting either ASEDs or normal saline eye drops;and 2 occurred after the Month 6 visit when participants had the option of continuing either ASEDs or normal saline eye drops
Groups:
- ASEDs: Adverse event occurred when participants were receiving autologous serum eye drops (ASEDs) daily during the crossover period (first six months) of the study.
- Saline: Adverse event occurred when participants were receiving control (normal saline) eye drops daily during the crossover period (first six months) of the study.
- ASEDs or Saline: Adverse event occurred after the Month 6 visit when participants had the option of continuing either ASEDs or normal saline eye drops daily if desired.
- No Intervention: Adverse event occurred prior to participants receiving either intervention. Neither ASEDs nor normal saline eye drops were being taken when the event occurred.
Arm/Group | ASEDs | Saline | ASEDs or Saline | No Intervention
Serious Adverse Events (participants affected / at risk) | 1/18 | 0/18 | 2/18 | 1/18
Other Adverse Events (participants affected / at risk) | 0/18 | 2/18 | 0/18 | 1/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ASEDs (N=18) | Saline (N=18) | ASEDs or Saline (N=18) | No Intervention (N=18)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspergillus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ASEDs (N=18) | Saline (N=18) | ASEDs or Saline (N=18) | No Intervention (N=18)
Retinal vein occlusion (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Macular oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract subcapsular (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes